CLINICAL TRIAL: NCT04888624
Title: A Comparison Between Two Post-operative Dressings in the Treatment of Surgical Incisions in Healthy Volunteers
Brief Title: A Comparison Between Two Post-operative Dressings
Acronym: DrySee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SerenaGroup, Inc. (Network)
Collaborators: DrySee, Inc (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DRYSEE-001
Record Dates: First submitted 2021-05-04; First posted 2021-05-17 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Surgical Incision
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Intervention Model Description: Healthy subjects drawn from the general population. will undergo a 1.5cm incision on the volar forearm of each arm. The incision will be closed with streriostrips. The subject's incisions will then be randomized to receive either a Tegaderm® + Pad transparent film dressing or DrySee® dressing with moisture detection. The incisions will be photographed three times per week. Data on dressing wear time, integrity and adverse events will be collected every two days in the clinic.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- DrySee® dressing with moisture detection (Experimental): DrySee® dressing with moisture detection
  Interventions: Device: DrySee® dressing with moisture detection
- Tegaderm® + Pad transparent film dressing (Active Comparator): Tegaderm® + Pad transparent film dressing
  Interventions: Device: Tegaderm® + Pad transparent film dressing

INTERVENTIONS:
Device: DrySee® dressing with moisture detection — DrySee® is a waterproof bandage designed to protect surgical incisions. It contains an indicator at the perimeter of the dressing, and at the wound site that turns blue when it comes into contact with liquid (figure 1). The indicator identifies a break in the integrity of the postoperative dressing. Changing the dressing at this point prevents bacteria from reaching the incision reducing the risk of infection. In addition, the waterproof dressing allows patients to shower or bath following surgery.
  Arms: DrySee® dressing with moisture detection
Device: Tegaderm® + Pad transparent film dressing — Tegaderm® is a transparent adhesive dressing commonly used as a postoperative dressing. The dressing has been shown to be superior to gauze in reducing SSIs. Tegaderm®, like DrySee,® is waterproof; however, it lacks technology that identifies a breach in dressing integrity.
  Arms: Tegaderm® + Pad transparent film dressing

SUMMARY:
Surgical site infections are one of the leading causes of post-operative morbidity and mortality worldwide. The ideal post-operative dressing is impermeable and remains intact preventing contamination of the incision with microorganisms. In addition, it is often difficult for the patient to identify breaks in dressing integrity. This trial compares a post-operative dressing (DrySee® Inc. Houston Tx) with moisture detection allowing the patient to recognize when the dressing is compromised to a standard post-operative dressing (Tegaderm® + Pad, 3M, St. Paul, MN). The ideal dressing also allows the patient to shower without removing the dressing.

DETAILED DESCRIPTION:
Healthy subjects drawn from the general population. will undergo a 1.5cm incision on the volar forearm of each arm. The incision will be closed with streriostrips. The subject's incisions will then be randomized to receive either a Tegaderm® + Pad transparent film dressing or DrySee® dressing with moisture detection. The incisions will be photographed three times per week. Data on dressing wear time, integrity and adverse events will be collected every two days in the clinic.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old.
2. Subject has read, understood, and signed approved consent, and is willing to participate and comply with the study procedures and requirements.

Exclusion Criteria:

1. Subject on an investigational drug or therapeutic device within 30 days of the study visit.
2. Presence of a condition that PI considers will compromise the subject's ability to participate in the study.
3. Known allergy to any of the dressings or their components.
4. The subject has a history of excessive bleeding.
5. The subject has a history of keloid formation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
A comparison of wear time between the two post-operative dressings under study. | 6-weeks
  A comparison of wear time between the two post-operative dressings under study.

SECONDARY OUTCOMES:
The effectiveness of liquid indication in identifying dressing compromise by visual assessment | 6-weeks
  The effectiveness of liquid indicator of the dressing turning blue
A comparison of dressing integrity between the two dressings under study if the dressings remains intact at the treatment visits by visual assessment. | 6-weeks
  A comparison of dressing integrity between the two dressings under study if the dressings remains intact at the treatment visits by visual assessment.
A comparison between the two dressings to maintain waterproof protection of the incision by visual assessment if there was a break in the dressing border. | 6-weeks
  A comparison between the two dressings to maintain waterproof protection of the incision by visual assessment of if there was a break in the dressing border at each treatment visit.
A comparison of adverse events between the two treatment arms. | 6-weeks
  A comparison of adverse events between the two treatment arms.

OTHER OUTCOMES:
A comparison of bacterial burden beneath the two dressings measured by fluorescence imaging (MolecuLight, Toronto, CA). | 6-weeks
  A comparison of bacterial burden beneath the two dressings measured by fluorescence imaging (MolecuLight, Toronto, CA).

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Serena, MD,FACS, Principal Investigator — SerenaGroup, Inc.
Locations (1):
- Serena Group Monroeville, Monroeville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No